CLINICAL TRIAL: NCT04507893
Title: Clinical, Laboratory and Imaging Comparison Between COVID-19 Pneumonia Confirmed by PCR Detection on Nasopharyngeal Swab and Negative Swab Pneumonia
Brief Title: Comparison Between Positive and Negative COVID-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Clinical Professor, University of Palermo
Other Study IDs: ACPM26
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Interstitial Pneumonia
MeSH Terms: conditions — COVID-19; Lung Diseases, Interstitial | interventions — Laboratories

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-COV-2 PNEUMONIA CONFIRMED BY PCR ON NASOPHARYNGEAL SWAB: Hospitalized patients affected by COVID-19 interstitial pneumonia (with positive PCR on naso-pharyngeal swab)
  Interventions: Other: Clinical, laboratory and imaging characteristics of pneumonia
- NEGATIVE SARS-COV-2 PNEUMONIA: Hospitalized patients affected by negative COVID-19 interstitial pneumonia (with negative PCR on naso-pharyngeal swab)
  Interventions: Other: Clinical, laboratory and imaging characteristics of pneumonia

INTERVENTIONS:
Other: Clinical, laboratory and imaging characteristics of pneumonia — Evaluation of the clinical, laboratory and imaging characteristics in patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay for COVID-19 on naso-pharyngeal swab as "COVID-19 patients" and "negative COVID-19 patients".

SUMMARY:
In the late 2019 a new Coronavirus was identified as the cause of a group of atypical interstitial pneumonia cases in Wuhan, a city in the Chinese province of Hubei. In February 2020, the World Health Organization designated COVID-19 disease, which stands for Coronavirus 2019 disease. Following the progressive spread of the infection in other countries of the world, WHO declared the Pandemic on 11 March 2020. Italy was the first European country involved in the spread of the infection and among those with the highest number of victims. The Coronavirus responsible for COVID-19 has, as its main target organ, the respiratory system, being able to determine a serious acute respiratory syndrome similar to that of the cases found during the SARS epidemic of 2003: hence the name of the virus as SARS-CoV-2. The diagnosis of SARS-COV-2 infection is made by direct detection by PCR of viral RNA on different biological materials from patients with suspicious symptoms, and the first level diagnostic test is generally the nasopharyngeal swab. However, even if the specificity of the nasopharyngeal swab is high, its sensitivity can be affected by technical causes (sampling mode), as well as by intrinsic factors related to the method. The purpose of the study is to identify the clinical, laboratory and imaging characteristic which are similar or which can differentiate the hospitalized patients affected by COVID-19 pneumonia (with positive PCR on naso-pharyngeal swab) and patients with pneumonia with negative PCR for COVID-19. To do this, the investigators will compare the clinical, laboratory and imaging characteristics between interstitial pneumonia secondary to SARS-COV-2 infection, confirmed by molecular biology investigations (viral RNA research by PCR on nasopharyngeal swab) and cases of interstitial pneumonia negative to the nasopharyngeal swab.

DETAILED DESCRIPTION:
In the late 2019 a new Coronavirus was identified as the cause of a group of atypical interstitial pneumonia cases in Wuhan, a city in the Chinese province of Hubei. In February 2020, the World Health Organization designated COVID-19 disease, which stands for Coronavirus 2019 disease. Following the progressive spread of the infection in other countries of the world, WHO declared the Pandemic on 11 March 2020. Italy was the first European country involved in the spread of the infection and among those with the highest number of victims. The Coronavirus responsible for COVID-19 has, as its main target organ, the respiratory system, being able to determine a serious acute respiratory syndrome similar to that of the cases found during the SARS epidemic of 2003: hence the name of the virus as SARS-CoV-2. Multisystem involvement and hyperinflammatory organ and systemic response are responsible for the patient's death. Overall, hospital mortality from COVID-19 is approximately 15% to 20%, but up to 40% among patients requiring ICU admission. The diagnosis of SARS-COV-2 infection is made by direct detection of viral RNA on different biological materials from patients with suspicious symptoms, and the first level diagnostic test is generally the nasopharyngeal swab; molecular investigations can also be carried out on samples from the distal respiratory tract (BronchoAlveolar Lavage, BAL). However, even if the specificity of the nasopharyngeal swab is high, its sensitivity can be affected by technical causes (sampling mode), as well as by intrinsic factors related to the method. The sensitivity data available are around 40-70%. The result is the possibility of a consistent series of false negatives (at least one third), represented by patients which have clinical characteristics compatible with SARS-COV-2 infection, but resulted, however, negative to the nasopharyngeal swab. These cases are framed as COVID-19-like cases and constitute a serious problem for the risk of not to recognize hospitalized patients suffering from COVID-19 infection.

The purpose of the study is to identify the clinical, laboratory and imaging characteristic which are similar or which can differentiate the hospitalized patients affected by COVID-19 pneumonia (with positive PCR on naso-pharyngeal swab) and patients with pneumonia with negative PCR for COVID-19. To do this, the investigators will compare the clinical, laboratory and imaging characteristics between interstitial pneumonia secondary to SARS-COV-2 infection, confirmed by molecular biology investigations (viral RNA research by PCR on nasopharyngeal swab) and cases of interstitial pneumonia negative to the nasopharyngeal swab. The cases studied will be represented by patients hospitalized for interstitial pneumonia in the participating hospital centers in the period between mid-March 2020 and end of May 2020. For these cases, all available data contained in the medical records of patients, enrolled within the time frame indicated above, will be retrospectively analyzed. Due to relative lack of sensitivity of COVID-19 PCR assay in nasopharyngeal swab, patients affected with COVID-19 infection can be mixed with other hospitalized patients and with unprotected health staff. On the basis of the comparison of the clinical, laboratory and imaging data the study would identify the characteristics which can differentiate patients with SARS-COV-2 pneumonia, confirmed by nasopharyngeal swab, and interstitial pneumonia and negative COVID-19 PCR on swab. The investigators aim to highlight any similarities or differences or the need for differentiated treatments.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients referred to the Emergency Unit of the "V. Cervello" Hospital, in Palermo, Italy, for clinical symptoms suggestive of suspected COVID-19 infection.

In details, we consider patients referred for one or more of the following manifestations: respiratory symptoms, fever, taste or smell loss.

To be included their records must include:

* detailed clinical history
* radiological findings (High-resolution CT, HRCT)
* results of viral RNA research for SARS-COV2, by PCR on nasopharyngeal swab, repeated two times (at the admission and again after 48 hours from the admission in the Emergency Unit)
* laboratory results regarding routine hemato-chemical assays
* oxygen therapy
* treatment used.

Exclusion Criteria:

* age <18 years
* incomplete medical records with respect to the parameters sought

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective, multicenter study, conducted on patients with interstitial pneumonia, admitted, consecutively, to the Internal Medicine I Unit of the "Villa Sofia - Cervello" Hospitals of Palermo, and two other Units dedicated to Patients affected with COVID-19, in the same hospital, from March 15, 2020 to May 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical characteristics of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Accuracy of severity of respiratory insufficiency - evaluated as need of three step "nasal oxygen, oxygen mask, invasive ventilation" - in differentiate COVID-19 infection, classified according to the results of PCR assay for COVID-19 on naso-pharyngeal swab as "COVID-19 patients" and "COVID-19 negative controls"
Evaluation of the laboratory characteristics of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Accuracy of the association of 3 haemato-chemical abnormalities (lymphopenia + increased serum transaminases + increased serum LDH) in differentiate COVID-19 infection, classified according to the results of PCR assay for COVID-19 on naso-pharyngeal swab as "COVID-19 patients" and "COVID-19 negative controls".
Evaluation of the imaging characteristics of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Accuracy of thorax CT scan in differentiate COVID-19 infection, classified according to the results of PCR assay for COVID-19 on naso-pharyngeal swab as "COVID-19 patients" and "COVID-19 negative controls".

SECONDARY OUTCOMES:
Evaluation of mortality of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Evaluation of mortality in "COVID-19 patients" and "COVID-19 negative controls", hospitalized in the study period.
Evaluation of clinical severity of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Evaluation of clinical severity in "COVID-19 patients" and "COVID-19 negative controls", hospitalized in the study period.
Evaluation of hospital stay length of patients with clinical presentation suggestive of COVID-19 infection, classified according to the results of PCR assay as "COVID-19 patients" and "COVID-19 negative controls". | 75 Days
  Evaluation of hospital stay length in "COVID-19 patients" and "COVID-19 negative controls", hospitalized in the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Principal Investigator — University of Palermo
Locations (3):
- Italy (3):
  - Infectious diseases Unit of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Pulmonology Unit Dedicated to COVID-19 Patients, Palermo, PA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Mitri C, Arcoleo G, Mazzuca E, Camarda G, Farinella EM, Soresi M, Carroccio A; IMUSG. COVID-19 and non-COVID-19 pneumonia: a comparison. Ann Med. 2021 Dec;53(1):2321-2331. doi: 10.1080/07853890.2021.2010797. PMID 34854790